CLINICAL TRIAL: NCT00623272
Title: Left Ventricular Function Assessment After Acute Myocardial Infarction: Comparison Between bi-, Three-dimensional and Cardiac Magnetic Resonance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007 28; 2007-A01081-52
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2008-06

CONDITIONS: Acute Myocardial Infarction
Keywords: The assessment of left ventricular ejection fraction (LVEF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: compare measurements of left ventricular volumes and LVEF (by Cardiac Magnetic Resonance and Echocardiography) — To compare measurements of left ventricular volumes and LVEF obtained by 2DE, 3DE, and CMR after a ST elevation myocardial infarction (STEMI) complicated by systolic left ventricular dysfunction.

SUMMARY:
compare measurements of left ventricular volumes and LVEF obtained by 2DE, 3DE, and CMR after a ST elevation myocardial infarction (STEMI) complicated by systolic left ventricular dysfunction

DETAILED DESCRIPTION:
The assessment of left ventricular ejection fraction (LVEF) is a critical step after a myocardial infarction because it determines the prognosis and the therapeutic management (indication of implantable cardioverter-defibrillators). Three-dimensional echocardiography (3DE) and cardiac magnetic resonance (CMR) are accurate and reproducible techniques to quantify left ventricular volumes and LVEF. However, all the large randomized trials which evaluated the role of the implantable cardioverter-defibrillators (ICD) on survival in primary prevention were based on LVEF values obtained by older techniques like bi-dimensional echocardiography (2DE), angiography or radionuclide scanning. From now, no study has compared the measurements of left ventricular volumes and LVEF obtained by further current techniques after an acute myocardial infarction (AMI) particularly after 1 month when ICD could be indicated.

ELIGIBILITY:
Inclusion Criteria:

* All the patients presenting a first ischemic clinical episode for at least 30 minutes, associated with one known gap will be included in a forward-looking and consecutive way, of at least 0.1mV in at least two peripheral diversions of the same territory or of at least 0.2 mV in at least two precordial diversions of the same territory
* An initial FEVG (measured by echocardiography or ventricular angiography in the daytime of the admittance)

Exclusion Criteria:

* Age < 18 years
* Antecedents of IDM
* Contraindications in the MRI (claustrophobia, stimulating and defibrillators heart patient implantable, metal intraocular brightness, allergy in the gadolinium, the severe renal insufficiency with clearance in the creatinine ≤30 mL/min)
* Fibrillation little finger
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
compare measurements of left ventricular volumes and LVEF obtained by 2DE, 3DE, and CMR after a ST elevation myocardial infarction (STEMI) complicated by systolic left ventricular dysfunction. | 3 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: franck THUNY, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Timone's hospital, Marseille, France